CLINICAL TRIAL: NCT03683407
Title: Effect of Platinum-based Chemotherapy on Tumor Mutation Burden in Patients With Advanced Non-small Cell Lung Cancer
Brief Title: Effect of Chemotherapy on TMB in NSCLC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Baodong Qin (Other)
Responsible Party: Sponsor-Investigator, Baodong Qin, Principal Investigator, Shanghai Changzheng Hospital
Organization: Shanghai Changzheng Hospital (Other)
Other Study IDs: COTMB
Record Dates: First submitted 2018-09-16; First posted 2018-09-25 (Actual); Last update posted 2018-09-25 (Actual); Status verified 2018-09

CONDITIONS: Chemotherapy Effect; Immunotherapy; Tumor Mutation Burden; PD-1/L1 Inhibitor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA from tumor tissue or circulating Tumor DNA
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chemotherapy Group: All participants are advanced NSCLC without druggable gene mutation (EGFR, ALK, ROS-1, Met, Ret. BRAF, etc), who would receive platinum-based chemotherapy.
  Interventions: Other: Next-Genernation Sequence

INTERVENTIONS:
Other: Next-Genernation Sequence — Tumor Mutation burden will be evaluated using NGS after 2-cycle chemotherapy, 4-cycle chemotherapy, or at progressive disease

SUMMARY:
Tumor mutation burden is identified as an important biomarkers for predicting PD-1/PD-L1 inhibitors in advanced Non-Small Cell Lung Cancer. Several previous clinical trials have demonstrated that chemotherapy could enhance the efficacy of PD-1/L1 immunotherapy in NSCLC such as Checkmate-227, Impower-150, Keynote-189, etc. Pre-clincial experiment shows that chemotherapy could increase CD8 TIL infiltration in tumor microenvironment, activate T cell immune reaction. However, it remains unclear whether chemotherapy could affect tumor mutation burden in advanced NSCLC patients. The present study aims to evaluate whether tumor mutation burden will change after receiving chemotherapy in advanced NSCLC patients.

ELIGIBILITY:
Inclusion Criteria:

* Advanced NSCLC diagnosed histologically; Expected survival ≥ 6 month;
* Without Druggable molecular events (EGFR, ALK, c-Met, BRAF, Ret, etc)
* ECOG / PS score: 0-2, and the main organ function to meet the following criteria: HB ≥ 90g / L, ANC ≥ 1.5 × 109 / L, PLT ≥ 80 × 109 / L,BIL <1.5 times the upper limit of normal (ULN); Liver ALT and AST <2.5 × ULN and if liver metastases, ALT and AST <5 × ULN; Serum Cr ≤ 1 × ULN, endogenous creatinine clearance ≥50ml/min

Exclusion Criteria:

* Patient can not comply with research program requirements or follow-up;
* Patient will receive immunotherapy;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Advanced NSCLC without druggable molecular events (EGFR, ALK, c-Met, BRAF, Ret, etc)
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-02-28 (Estimated); Study Completion 2019-08-31 (Estimated)

PRIMARY OUTCOMES:
Tumor Mutation Burden Change | every 6 weeks up to progression disease
  Tumor mutation burden will be calculated using a 520 genes NGS panel

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No